CLINICAL TRIAL: NCT02965846
Title: Topical Ophthalmic AGN-195263 for the Treatment of Evaporative Dry Eye
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 195263-010
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Results first posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Dry Eye Syndromes
Keywords: EDE; evaporative dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AGN-195263 (Experimental)
  Interventions: Drug: AGN-195263
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: AGN-195263 — 1 drop of AGN-195263 will be instilled in each eye twice daily.
  Arms: AGN-195263
Drug: Vehicle — 1 drop of AGN-195263 vehicle(placebo) will be instilled in each eye twice daily.
  Arms: Vehicle

SUMMARY:
The objectives of this study are twofold •To evaluate the safety and efficacy of 0.1% AGN-195263 administered twice daily compared to its vehicle in patients with evaporative dry eye (EDE) •To evaluate the systemic pharmacokinetics of 0.1% AGN-195263 administered twice daily in patients with EDE

ELIGIBILITY:
Inclusion Criteria:

* Male, 18 years of age or older, at the screening (day -51) visit OR
* Females, who are naturally postmenopausal (permanent cessation of menstrual periods for at least 12 consecutive months) or are permanently sterilized (ie, eg, tubal occlusion,hysterectomy, bilateral salpingectomy, and/or bilateral oophorectomy) at the screening (day -51) visit
* In at least 1 eye, all of the following objective measures of evaporative dry eye (EDE) must be present at the standardization (day -21) and baseline (day 1) visits. The same eye must qualify at both visits

  * Tear film break-up time (TBUT) ≥ 2 seconds and ≤ 7 seconds
  * Corneal sodium fluorescein staining score ≥ 1 and ≤ 4 (Oxford scheme)
  * Anesthetized Schirmer's tear test score ≥ 10 mm after 5 minutes
* At the standardization (day -21) and baseline (day 1) visits, patients must have:

  * Ocular Surface Disease Index© (OSDI) score > 12 (0 to 100 scale)
  * Overall ocular discomfort score ≥ 1 and < 4 (0 to 4 scale; 0 = none, 4 = very severe)
  * Ocular burning score ≥ 1 and < 4 (0 to 4 scale; 0 = none, 4 = very severe)
  * Blurred vision score ≥ 1 and < 4 (0 to 4 scale; 0 = none, 4 = very severe)
* In at least 1 eye, a lower lid margin meibum quality global assessment score ≥ 1 at the standardization (day -21) and baseline (day 1) visits. The same eye must qualify at both visits
* In at least 1 eye, the number of lower lid margin expressible meibomian glands must be ≥ 3 at the standardization (day -21) and baseline (day 1) visits. The same eye must qualify at both visits
* Use of an artificial tear product, lid hygiene (ie, warm compress, lid massage, lid scrub), omega-3 supplementation (topical ocular or systemic), or antibiotics (ie, systemic or topical macrolides, tetracyclines, tetracycline derivatives [including doxycycline and minocycline]) for the treatment of dry eye disease, or meibomian gland disease within 1 year of the standardization (day -21) visit

Exclusion Criteria:

* Male patients with a history of, known, or suspected prostate cancer
* Male patients with a prostate-specific antigen (PSA) level ≥ 4 μg/L
* Female patients with a history of known or suspected breast, cervical, ovarian, or uterine cancer
* Female patient who is of child-bearing potential
* At standardization (day -21) and / or baseline (day 1) visits, a lower lid margin meibum quality global assessment score of non-expressible (NE) in either eye
* Patients who are currently using estrogen and/or progesterone containing products (including herbal and nutritional supplements) and not on a stable dose (at least 90 days prior to the standardization visit (day -21) and/or anticipate initiating use and/or changing use during the study
* Patients who are currently using or have used any androgen or anti-androgen treatment (including herbal and nutritional supplements), within 90 days of the standardization (day -21) visit or anticipated use during the study
* Patients who are currently using or have used any hair growth product within 90 days of the standardization (day -21) visit or anticipated use during the study
* Patients who are currently using or have used topical corticosteroids in the eyes or on the eyelids within 60 days prior to the standardization visit (day -21), or any such use anticipated prior to the month 6 visit
* Patients who are currently using or have used oral or topical macrolides, tetracyclines, tetracycline derivative drugs (including doxycycline and minocycline), retinoids (eg, isotretinoin), calcineurin inhibitors (ie, RESTASIS®, Ikervis®), oral (systemic) corticosteroids, or lifitegrast (Xiidra™) or any other therapeutic dry eye treatment within 60 days of the standardization visit (day -21), or anticipated use before the month 6 visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2017-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khristopher Hansen, Study Director — Allergan
Locations (49):
- United States (8):
  - Sall Research Medical Center, Artesia, California
  - Lugene Eye Institute, Glendale, California
  - Lifelong Vision Foundation, Chesterfield, Missouri
  - Devers Eye Institute, Portland, Oregon
  - Scott and Christie Associates, Cranberry Township, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Piedmont Eye Center, Lynchburg, Virginia
- Czechia (4):
  - Fakultni nemocnice Ostrava, Ostrava
  - Ocni klinika OFTEX, Pardubice
  - FN Kralovske Vinohrady, Ocni Klinika, Prague
  - Oční ambulance, Velká Bíteš
- France (3):
  - CHU de Bordeaux, Service d'Ophtalmologie, Bordeaux
  - CHU Hopital Morvan (Bat 4) Service Daviel Ophtalmologie, Brest
  - CHU Limoges - Hôpital Dupuytren, Limoges
- Germany (6):
  - University Hospital of Cologne, Dept of Ophthalmology, Cologne
  - Augenklinik Universitatsklinikum, Düsseldorf
  - University Eye Hospital, Freiburg im Breisgau
  - Gutenberg University Medical School, Dept of Ophthalmology, Mainz
  - Ludwig-Maximilians-University, Dept of Ophthalmology, Munich
  - St. Franziskus Hospital Augenabteilung, Münster
- Hungary (3):
  - Dept. of Ophthalmology Semmelweis University, Budapest
  - University of Debrecen, Dept of Opthalmology, (DE OEC Szemklinika), Debrecen
  - University of Szeged Szent-Györgyi Albert Clinical Center, Faculty of Medicine, Dept of Ophthalmology, Szeged
- Italy (5):
  - Rapallo Hospital, Opthalmology Department, Genova
  - Istituto di Oftalmologia, Messina
  - Ospedale San Giuseppe, Universita di Milano, Milan
  - Istituto Di Ricovero E Cura A Carattere Scientifico (IRCCS) - Ospedale San Raffaele (HSR) (Istituto Scientifico Universitario San Raffaele), Milan
  - University of Pisa, Neurosciences - Section of Ophthalmology, Pisa
- Philippines (3):
  - Asian Eye Institute, Makati City
  - Peregrine Eye and Laser Institute, Makati City
  - The Medical City, Pasig
- Poland (5):
  - Prywatna Klinika Okulistyczna OFTALMIKA, Bydgoszcz
  - Szpital Specjalistyczny nr 1 w Bytomiu, Bytom
  - Optimum Profesorskie Centrum Okulistyki, Gdansk
  - Specjalistyczna Praktyka Lekarska prof. Edward Wylegala, Katowice
  - Uniwersyteck Szpital Kliniczny im. Jana Mikulicza-Radeckiego, Wroclaw
- Spain (6):
  - Institto de Microcirugia Ocular C/Josep Maria Llado, Barcelona
  - Clinico de Barcelona Casa de la Maternidad, Barcelona
  - Clinica Oftalmologica, Huelva
  - Instituto Oftalmologico Fernandez-Vega, Oviedo, Principado de Asturias
  - Cartuja Vision, Seville
  - University of Valladolid, Facultad Medicina, Valladolid
- Taiwan (3):
  - Buddhist Tzu Chi General Hospital, Hualien City
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- Turkey (Türkiye) (2):
  - Ege Üniv. Tıp Fakültesi, Izmir
  - Erciyes Üniversitesi Tıp Fakültesi, Kayseri
- Newcastle University School of Medicine, Dept of Ophthamology, Newcastle upon Tyne, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 43 participants who enrolled in the study, 10 were randomized and received intervention to compromise the safety and Intent to Treat (ITT) populations
Groups:
- AGN-195263: One drop of 0.1% AGN-195263 instilled in each eye twice daily
- Vehicle: One drop of Vehicle (placebo) instilled in each eye twice daily
- Enrolled But Not Randomized: Run-In period before randomization
Period: Overall Study
Arm/Group | AGN-195263 | Vehicle | Enrolled But Not Randomized
Started | 5 | 5 | 33
Completed | 0 | 0 | 0
Not Completed | 5 | 5 | 33
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Study Terminated By Sponsor | 4 | 4 | 0
Not completed — Participants not randomized | 0 | 0 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN-195263 | Vehicle | Enrolled But Not Randomized | Total
Number analyzed (Participants) | 5 | 5 | 33 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 27 | 36
  >=65 years | 0 | 1 | 6 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 23 | 26
  Male | 3 | 4 | 10 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 6 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 3 | 4 | 10 | 17
  White | 2 | 1 | 16 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index Population: Data missing for 8 out of the 33 participants in the enrolled but not randomized arm.
  kg/m^2
    number analyzed (Participants) | 5 | 5 | 25 | 35
    (all) | 34.34 (10.649807509998) | 34.86 (9.1331484166195) | 32.788 (9.4405643899081) | 33.996 (.65464394984732)
Weight [Mean (Standard Deviation); unit: kg] — Population: Data missing for 8 out of the 33 participants in the enrolled but not randomized arm.
  kg
    number analyzed (Participants) | 5 | 5 | 25 | 35
    (all) | 101.44 (23.543542639119) | 102.56 (20.180247768548) | 87.868 (25.016006395906) | 97.2893 (2.0238704230461)
Height [Mean (Standard Deviation); unit: cm] — Population: Data missing for 8 out of the 33 participants in the enrolled but not randomized arm.
  cm
    number analyzed (Participants) | 5 | 5 | 25 | 35
    (all) | 173.44 (5.6683683719391) | 172.9 (5.8343808583259) | 163.74 (9.2099077085495) | 170.026 (1.6317762147419)

OUTCOME MEASURES:

1. Primary Outcome: Overall Ocular Discomfort Score (0 to 4 Scale; 0=None, 4=Very Severe)
Description: The overall ocular discomfort will be assessed on a questionnaire using a 0 to 4 scale on which 0=none, 1=mild, 2=moderate, 3=severe and 4=very severe.
Time Frame: 6 month visit
Population: Efficacy analyses including the overall ocular discomfort score were planned. Ultimately, these analyses were not performed due to the fact that the study was terminated before the primary/secondary efficacy visit could be reached.
Arm/Group | AGN-195263 | Vehicle
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in Tearfilm Break Up Time (TBUT)
Description: For TBUT, the mean of 3 measurements of time in seconds will be computed at each visit for each eye. The mean value of the study eye will be used for the analysis.
Time Frame: Baseline (day 1) to 6 month visit
Population: Efficacy analyses including the change from baseline in Tearfilm Break Up Time (TBUT) were planned. Ultimately, these analyses were not performed due to the fact that the study was terminated before the primary/secondary efficacy visit could be reached.
Arm/Group | AGN-195263 | Vehicle
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 157 days
Description: Adverse Events were collected for randomized patients only.
Arm/Group | AGN-195263 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 1/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AGN-195263 (N=5) | Vehicle (N=5)
Vision Blurred (Eye disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to study termination, the study was underpowered

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As this study was terminated, no data will be published.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT02965846/Prot_SAP_000.pdf